CLINICAL TRIAL: NCT04043910
Title: Functional Near Infra-Red Spectroscopic Study of Central Auditory System Cortical Functional Reorganization in Unilateral Deaf Children
Brief Title: Functional Near Infra-Red Spectroscopic Study of Central Auditory System Cortical Functional Reorganization
Acronym: SUN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very difficult to include all patients
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0321
Record Dates: First submitted 2019-05-27; First posted 2019-08-02 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Hearing Loss, Unilateral
Keywords: Functional Neuroimaging; Pediatrics; fNIRS; Single-sided deafness
MeSH Terms: conditions — Hearing Loss, Unilateral | interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-sided deaf group (Experimental): 30 children will be included in this group
  Interventions: Device: fNIRS; Other: Speech intelligibility; Other: Sound localisation; Other: Speech assessments; Other: Quality of Life
- Normal hearing group (Active Comparator): 30 children will be included in this group
  Interventions: Device: fNIRS; Other: Speech intelligibility; Other: Sound localisation; Other: Speech assessments; Other: Quality of Life

INTERVENTIONS:
Device: fNIRS — The auditory cortical imaging will be performed by fNIRS measures. This non-invasive functional imaging technique relies on the use of a sensor-bearing cap, measuring cortical activity through scalp, during auditory stimulation. As head movement does not alter measurement that much, fNIRS is well adapted to children.
Other: Speech intelligibility — Speech intelligibility will be evaluated with French sentences comprehension in noise, from the Common Test or Adaptive Auditive Speech Test before 6 years, from the Common Test or Hearing in Noise Test for Children (Hint-C) from 7 to 11 years, and from the Hint-C or Marginal Benefit of Acoustic Amplification after 11 years, both with a Signal over Noise Ratio of +10 decibel at 65 decibel
Other: Sound localisation — Sound localisation will be evaluated with a left-right discrimination test before 7 years and a 12 loudspeakers sound localisation test after 7 years.
Other: Speech assessments — Speech assessments will be performed by dedicated speech therapists, with child age specific tests, and 2 global speech scores: the Category of Auditory Performances scale - second edition, and the Speech Intelligibility Rating scale.
Other: Quality of Life — Quality of Life (QoL) evaluation will be based on the generic QoL scale, and the Speech Spatial and Qualities of hearing (SSQ) deafness specific scale. Each scale exists in age specific modalities.

SUMMARY:
This study aims to compare the auditory cortical activity in response to monaural and binaural stimuli, measured by functional Near-Infrared Spectroscopy (fNIRS) between Single-sided Deaf (SSD) Children, and Normal-Hearing (NH) children from 5 to 16 years. Binaural audiological performance, speech skills and quality of life (QoL) will be compared between the 2 groups and links to with the cortical activity will be assessed.

DETAILED DESCRIPTION:
Binaural hearing allows strengthening of speech intelligibility in noise and sound localization. It is well known that single-sided (SSD) and bilateral asymmetric deafness lead to socio-behavioral consequences and, in children, inducing impairments in learning acquisitions.

In adults, SSD is associated with a reduction of inter-hemispheric functional asymmetry of auditory cortex on functional Magnetic Resonance Imaging. Moreover, in children with bilateral profound deafness who got one cochlear implant (inducing a form of asymmetric hearing), these clinical and functional anomalies cannot be overcome in case of a late (>1,5year) secondary implantation. This shows that once the loss of asymmetry is installed, it is difficult to recover from it.

No data about SSD in children and its cortical representation exists. In this study, the investigators hypothesized that SSD modifies the auditory cortical activation profile, linked with a deterioration of the binaural auditory skills, the global development and the quality of life If this hypothesis is confirmed, systematic and individualized rehabilitation will be needed to reduce patient's handicap and to prevent long term consequences.

The investigators will then measure the auditory cortical activity using fNIRS in 5 to 16 year-old SSD and NH children. The fNIRS system will use a sensor-bearing cap, measuring cortical activity through the scalp. Binaural hearing (speech in noise and localisation), speech assessments (global and speech development), and QoL will also be measured.

Children will undergo 2 sessions of 1 to 2 hours tests, each spaced up to 3 months apart. As they are children regularly seen in our ear-nose-throat department, a once-a-year follow-up will be proposed, on the child and his family convenience. As it is a non-interventional study, no follow-up would be needed.

ELIGIBILITY:
Inclusion Criteria :

For both groups:

* 5 to 16 year-old children,
* Absence of pregnancy
* Affiliation to Social Security, and children and their parents signed consents will be necessary.
* Participation agreement of the protocol and signature of the consent form by the person having parental authority and the child

For Single-sided Deafness subjects:

- shall present with moderate to profound unilateral hearing loss, with a hearing loss of 40 decibel(minimal thresholds), assessed on tonal, vocal audiometry, Auditory Brainstem Responses,

For Normal hearing subjects:

- shall have normal hearing, demonstrated by air thresholds below 20 decibel by an audiometric control before inclusion , matched in gender and age to children in the experimental group

Exclusion Criteria:

For both groups:

* Antecedents of Psycho-neurological diseases,
* Other sensorineural or motor deficiency,
* Familial bilingualism,
* Medications affecting vigilance.
* pregnancy or breastfeeding

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Oxyhemoglobin rates | 3 months
  Oxyhemoglobin (O2Hb) rates measured on the auditory cortex of each cerebral hemisphere during an auditory stimulus.
Deoxyhemoglobin rates | 3 months
  Deoxyhemoglobin (HHb) rates measured on the auditory cortex of each cerebral hemisphere during an auditory stimulus.

SECONDARY OUTCOMES:
Binaural audiological performances | 3 months
  Speech in noise intelligibility and spatial sound localization ability
Speech assessment | 3 months
  Hearing perception thanks to Category of Auditory Performances - Nottingham Early Assessment Package 4 and speech intelligibility thanks to the Speech Intelligibility Rating - Nottingham Early Assessment Package 5
Quality of life scores | 3 months
  Quality of Life (QoL) evaluation will be based on the KindLR generic QoL scale. This scale exists in age specific modalities.
Quality of life scores | 3 months
  Quality of Life (QoL) evaluation will be based on scale, and the Speech Spatial and Qualities of hearing (SSQ) deafness specific scale. This scale exists in age specific modalities.
Activity levels | 3 months
  fNIRS measured cortical of activity levels

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Noëlle CAMELS, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital Pierre Paul Riquet, Toulouse, France